CLINICAL TRIAL: NCT05784649
Title: Effects of Health Education Programs on Maternal Health Literacy, Health-promoting Behaviors and Empowerment of Rural Pregnant Women in China
Brief Title: Effects of Health Education Programs on the Health of Rural Pregnant Women in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20230228
Record Dates: First submitted 2023-02-28; First posted 2023-03-27 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Health Literacy
Keywords: health literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Other): The interventions of the control group will receive the routine health education proposed by relevant experts in China which are chosen by the Chinese Medical Association.
  Interventions: Other: health education
- intervention group (Experimental): The interventions of the intervention group will include routine health education. And then the participants will have individual counsel about health-promoting behaviors with a midwife and a doctor. The counseling will be based on the procedure of the health promotion model.
  Interventions: Behavioral: individual counsel

INTERVENTIONS:
Other: health education — The health education program will be conducted on the WeChat platform. The contents of health education include 1) knowledge about how to prevent anemia during pregnancy; 2) self-care education videos such as breastfeeding; 3) online courses on how to manage weight during pregnancy, and how to keep good emotions, etc.; 4) Nutrition and lifestyle guidance; 5) knowledge about recognition and prevention of risk factors or diseases: abortion, toxic substances, premature birth. The contents of health education will be totally shared 5 times from 12 weeks to 36 weeks in the pregnancy and once a month on the platform. Every participant should reply "read" after learning the contents. if they have any questions, they can reply for "help" for further connection with health professionals.
  Arms: control group
Behavioral: individual counsel — The participants will receive the same health education as the control group. The pregnant women will have one routine checkup a month from 12 weeks to 36 weeks in the hospital. And they will receive counseling with a midwife and a doctor after every routine checkup. The counseling will have a total of 5 times and once a month, 45 minutes per time. The professionals will evaluate health-promoting behaviors such as nutrition and physical activity based on the procedure of the health promotion model. The model includes four continued parts: prior behaviors; personal influences; interpersonal Influences; commitment to a plan of action. Finally, the professionals will give person-centered advice to help the participants practice the content of health education, keep health-promoting behaviors, and achieve a healthy lifestyle.
  Arms: intervention group

SUMMARY:
The aim of this study is to design, introduce, conduct, and evaluate health education programs to improve maternal health literacy, health-promoting behaviors, and empowerment of pregnant women in China.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, the quasi-experimental study will be conducted. All the pregnant women who meet the inclusion criteria will be marked as numbers in the first inspection time of the second trimester. And then the odd number will be assigned to an intervention group, while the even number will be distributed to the control group which ensures that they have an equal chance of receiving the intervention.The interventions of the control group will receive the routine health education proposed by relevant experts in China which are chosen by the Chinse Medical Association. The interventions of the intervention group will receive routine health education and individual counsel on health-promoting behaviours based on the health promotion model .

ELIGIBILITY:
Inclusion Criteria:

1. Adult pregnant women;
2. Basic reading and comprehension skills;
3. Can use WeChat app;
4. Can complete all evaluations;
5. Willing to receive guidance and change.
6. The home address shown on the identification card is in a rural area.

Exclusion Criteria:

1. Threatened abortion;
2. Premature rupture of membranes;
3. Serious complication;
4. Be absent from health education more than 2 times;
5. Have psychic or mental problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2024-05-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline scores of maternal health literacy at 3 months and 5 months | The changes in the scores will be evaluated before the first month (6 to 13+6 weeks), after 3 months (25 to 28 weeks), and 5 months (33 to 36 weeks) of the intervention.
  The health literacy scale for perinatal pregnant women was used to measure the level of maternal health literacy among Chinese pregnant women.It consists of 55 items accompanied by a 5-point Likert scale. The option of forward scoring items ranges from 5= strongly agree, 4 = agree, 3= uncertain, 2 = not agree, and 1 = strongly not agree. The option of reversed rescoring items ranges from 1= strongly agree, 2 = agree, 3= uncertain, 4 = not agree, and 5 = strongly not agree. The score is collected by calculating the participant's responses that form the total score from 51 to 255. The eligibility criteria were the ratio of personal score over total score is over 80% (204 points) .Based on the previous studies, the outcomes of similar interventions were tested before the first implementation of the intervention, at three months, and at the end of the intervention.
Change from Baseline scores of health-promoting behaviors at 3 months and 5 months | The changes in the scores will be evaluated before the first month (6 to 13+6 weeks), after 3 months (25 to 28 weeks), and 5 months (33 to 36 weeks) of the intervention.
  Health Promotion Lifestyle Profile-II (HPLP-II) was widely chosen to evaluate the health behaviors of pregnant women. The Chinese version of HPLP-II was formed with 40 items with scores ranging from 1 to 4. The total scores range from 40 to 160. The higher scores , the better health-promoting behaviors.Based on the previous studies, the outcomes of similar interventions were tested before the first implementation of the intervention, at three months, and at the end of the intervention.

SECONDARY OUTCOMES:
Change from Baseline scores of empowerment at 3 months and 5 months | The changes in the scores will be evaluated before the first month (6 to 13+6 weeks), after 3 months (25 to 28 weeks), and 5 months (33 to 36 weeks) of the intervention.
  The Empowerment Scale for Pregnant Women was used to evaluate the empowerment of pregnant women. This scale consists of 27 items with scores ranging from 1 to 4. The total scores range from 27 to 108. The higher scores, the better empowerment. Based on the previous studies, the outcomes of similar interventions were tested before the first implementation of the intervention, at three months, and at the end of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mei Chan Chong, Dr., Study Chair — univerisiti malaya; Yanjia Liu, Dr., Principal Investigator — universiti malaya
Locations (1):
- Faculty of medicine, Kuala Lumpur, None Selected, Malaysia

IPD SHARING:
Plan to Share IPD: No